CLINICAL TRIAL: NCT06256549
Title: A Multicenter, Randomized, Controlled Phase II Clinical Trial to Evaluate the Efficacy and Safety of GZR18 Injection in Chinese Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of GZR18 Injection in Chinese Patients With Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gan and Lee Pharmaceuticals, USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GL-GLP-CH2004
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GZR18 (Experimental): GZR18 injection s.c.
  Interventions: Drug: GZR18
- Semaglutide (Active Comparator): Semaglutide injection s.c.
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: GZR18 — Titrated to low dose or middle or high dose
  Arms: GZR18
Drug: Semaglutide — Titrated to 1.0 mg once a week
  Arms: Semaglutide

SUMMARY:
This study was a multicenter, randomized, parallel and controlled study in adult patients with T2DM to evaluate the efficacy, safety (including immunogenicity) and pharmacokinetics of GZR18 injection in adult patients with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* (1) Chinese adults, male or female aged between 18 and 75 (including both ends).

  (2) According to the diagnostic and classification criteria of diabetes issued by the World Health Organization (WHO) in 1999, and the supplementary diagnostic criteria of WHO in 2011, type 2 diabetes was diagnosed for more than 3 months.

  (3) Lifestyle intervention and / or unregulated use of antidiabetic drugs within 3 months before screening, or stable use of less than 3 oral hypoglycemic drugs within 3 months before screening.

  (4) HbA1c (HbA1c) ≥ 7.0% and ≤ 11% during screening.

  (5) Body mass index (BMI) ≥ 18.5 kg/m2.

  (6) There is no birth plan within 6 months from the signing of informed consent to the last administration, and those who voluntarily take effective contraceptive measures and have no sperm donation plan. Fertile women are not breastfeeding, and the screening and baseline pregnancy tests must be negative.

  (7) Patients fully understand the purpose, nature, methods and possible adverse reactions of the trial, can communicate well with researchers, and can understand and comply with the requirements of this study. During the study, they can maintain a stable diet and exercise lifestyle, and voluntarily sign an informed consent form to enter this study.

Exclusion Criteria:

* (1) Known or suspected to be allergic to GLP-1 drugs or their excipients, or have contraindications to their use.

  (2) Those who participated in clinical trials of other drugs or devices within 3 months before were screened and given treatment.

  (3) Surgery that can lead to weight instability was performed within 2 months before screening, or non-diabetic drugs that affect weight are currently being used or are in the weight loss program and are not in the maintenance stage.

  (4) History of alcohol or drug abuse, or positive results of pre-random drug abuse screening (urine screening).

  (5) Continuous use of insulin for more than 14 days in one year before screening (the time for gestational diabetes to receive insulin treatment is not within this limit); GLP-1RA drugs were used in the first 6 months; dipeptidyl peptidase-4 (DPP-4) inhibitors were used in the first month.

  (6) Growth hormone and other drug treatments determined by researchers to affect insulin levels were performed within 3 months before screening.

  (7) Diabetic ketoacidosis, diabetic lactic acidosis or hyperosmotic nonketotic diabetic coma within 6 months before screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2023-08-09 (Actual); Primary Completion 2024-07-20 (Estimated); Study Completion 2024-07-20 (Estimated)

PRIMARY OUTCOMES:
Compared with Semaglutide, the changes of HbA1c compared with baseline after continuous administration of GZR18 injection for 24 weeks | 24 weeks

SECONDARY OUTCOMES:
HbA1c compliance rate (< 7.0% and ≤ 6.5% of patients) | 24 weeks
  Compared with Semaglutide injection, GZR18 injection after continuous administration for 24 weeks
The overall incidence of adverse events and the incidence of serious adverse events | 27 weeks
  Compared with Semaglutide injection, GZR18 injection after continuous administration for 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Liyuan Zhao, Ph.D, Study Director — Gan & Lee Pharmaceuticals.
Locations (1):
- Gan & Lee Pharmaceuticals Co., Ltd, Beijing, China